CLINICAL TRIAL: NCT01089179
Title: An Open-Label, Randomized, 2-Period, 2-Treatment, Crossover, Single-Dose Bioequivalence Study of Metformin Hydrochloride Extended Release 500 mg Tablet (Test Formulation, Torrent Pharmaceuticals Ltd., India) Versus Glucophage XR® 500 mg Tablet (Reference Formulation, Bristol-Myers Squibb Company, USA) in Healthy Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Metformin Hydrochloride Extended Release 500 mg Tablet Versus Glucophage XR® 500 mg Tablet in Healthy Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: PK-07- 017
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Torrent's Metformin tablets 500 mg (Experimental)
  Interventions: Drug: Metformin
- Glucophage XR® of Bristol- Myers Squibb Company, USA) (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Objective: An Open-Label, Randomized, 2-Period, 2-Treatment, Crossover, Single- Dose Bioequivalence Study of Metformin Hydrochloride Extended Release 500 mg Tablet (Test formulation, Torrent Pharmaceuticals Ltd., India) Versus Glucophage XR® 500 mg Tablet (Reference formulation, Bristol- Myers Squibb company, USA) in Healthy Volunteers under Fed Conditions.

Study Design: An Open-Label, Randomised, 2-Period, 2-Treatment, Crossover Study under fed condition.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who qualify for the study should meet the following inclusion criteria.

  1. Male subjects in the range of 18 - 45 years of age.
  2. Body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart.
  3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and body temperature)
  4. Subjects with normal findings as determined by hematological tests, serum chemistry, urine analysis, ECG and X-ray.
  5. Willingness to follow the protocol requirement as evidenced by written, informed consent.
  6. Agreeing to, not using any medication (prescription and over the counter), including vitamins and minerals for two weeks prior to study & during the course of the study.
  7. No history or presence of significant alcoholism or drug abuse in the past one year.
  8. Non-smokers, ex smokers and light smokers will be included. " Light smokers are defined as someone smoking 10 cigarettes or less per day, ex smokers as someone who completely stopped smoking for at least 3 months.

Exclusion Criteria:

* The subjects who qualify for the study should not meet the following exclusion criteria:

  1. Requiring medication for any ailment including enzyme-modifying drugs Use of any drugs known to induce or inhibit hepatic drug metabolism (e.g.s, inducers: barbiturates, carbazepine, phenytoin, glucocorticoids, omeprazole; inhibitors: selective serotonin reuptake inhibitors (SSRIs), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
  2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
  3. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic or psychiatric diseases.
  4. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
  5. History of malignancy or other serious diseases.
  6. Refusal to abstain from food for ten (10) hours prior to study drug administration on first day of each study period and for four (4) additional hours each, post dose.
  7. Refusal to abstain from water for one hour pre dose and for two (2) hours, post dosing.
  8. Any contraindication to blood sampling.
  9. Refusal to abstain from smoking or consumption of tobacco products 24 hours before dosing until last sample collection of each period. Habituation of tobacco necessitating uninterrupted tobacco consumption.
  10. Use of xanthine-containing beverages or food for 48 hours prior to each drug dose.
  11. Blood donation 90 days prior to the commencement of the study.
  12. Subjects with positive HIV tests, HbsAg or Hepatitis-C tests.
  13. Known history of allergic reactions to Metformin or other related drugs.
  14. History of drug abuse in the past one year.
  15. Use of prescription medication or over the counter products (including natural food supplements,vitamins, garlic as a supplement) within 2 weeks prior to administration of study medication, except for topical products without systemic absorption.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Torrent Research Centre, Bhat, Gujarat, India

REFERENCES:
- See also: Related Info — http://www.fda.gov/